CLINICAL TRIAL: NCT00112736
Title: Phase I/II Study of OSI-774 (Erlotinib) and CCI-779 (Temsirolimus) in Patients With Recurrent Malignant Glioma
Brief Title: Erlotinib and Temsirolimus in Treating Patients With Recurrent Malignant Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02921; NCI-2012-02921 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000429553; NABTC04-02 (Other: Adult Brain Tumor Consortium); NABTC-04-02 (Other: CTEP); U01CA062399 (NIH); NCT00267878 (obsolete NCT alias)
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Results first posted 2015-06-15 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-05

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Oligodendroglioma; Adult Diffuse Astrocytoma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Mixed Glioma; Adult Pilocytic Astrocytoma; Adult Pineal Gland Astrocytoma; Adult Subependymal Giant Cell Astrocytoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Glioma; Brain Neoplasms | interventions — Erlotinib Hydrochloride; temsirolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase 1 (erlotinib & temsirolimus) (Experimental): PHASE I: Oral erlotinib 1 daily days 1-28 (150mg), temsirolimus IV 30 minutes days 1, 8, 15, 22 (dose escalation). Every 28 days until disease progression or unacceptable toxicity.
  pharmacological study: Correlative studies
  Interventions: Drug: erlotinib; Drug: temsirolimus; Other: pharmacological study
- Phase 2 temsirolimus MTD & erlotinib (Experimental): Oral erlotinib 1 daily days 1-28 (150mg), temsirolimus IV 30 minutes days 1, 8, 15, 22 at MTD phse I. Every 28 days until disease progression or unacceptable toxicity.
  PHASE II (preoperative component): Patients who are surgical candidates may opt to undergo surgical resection of the tumor. Beginning 5-7 days before surgery, these patients receive oral erlotinib once daily until surgery. Patients also receive temsirolimus IV over 30 minutes at the MTD and then undergo surgical resection of the tumor 3-24 hours later. Beginning 2-4 weeks after surgery, patients receive temsirolimus at the MTD and erlotinib as in phase I.
  therapeutic conventional surgery: Undergo surgical resection
  laboratory biomarker analysis: Correlative studies
  Interventions: Drug: erlotinib; Drug: temsirolimus; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: erlotinib — Given orally
  Other Names: CP-358,774; erlotinib hydrochloride; OSI-774
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel
Procedure: therapeutic conventional surgery — Undergo surgical resection
  Arms: Phase 2 temsirolimus MTD & erlotinib
Other: laboratory biomarker analysis — Correlative studies
  Arms: Phase 2 temsirolimus MTD & erlotinib
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
  Arms: Phase 1 (erlotinib & temsirolimus)

SUMMARY:
Erlotinib and temsirolimus and may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. This phase I/II trial is studying the side effects and best dose of temsirolimus when given together with erlotinib and to see how well they work in treating patients with recurrent malignant glioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the maximum tolerated dose (MTD) of OSI-774 (erlotinib; Tarceva) in combination with CCI-779 (temsirolimus) in patients with recurrent malignant glioma who are not taking enzyme-inducing anti-epileptic drugs (EIAEDs). (Phase I) II. To characterize the safety profile of OSI-774 (erlotinib) and CCI-779 (temsirolimus). (Phase I) III. To characterize the pharmacokinetics of OSI-774 (erlotinib) and CCI-779 (temsirolimus). (Phase I) IV. To determine the efficacy of OSI-774 (erlotinib) and CCI-779 (temsirolimus) in patients with recurrent malignant glioma as measured by 6-month progression-free survival. (Phase II)

SECONDARY OBJECTIVES:

I. Overall progression-free survival. (Phase II) II. Response. (Phase II)

TERTIARY OBJECTIVES:

I. To explore the association of response to treatment to the molecular phenotype of the tumor. (Phase II) II. Determine whether OSI-774 (erlotinib) and CCI-779 (temsirolimus) inhibits EGFR and mTOR and the PI3K-AKT-mTOR and RAS-ERK signaling pathways in tumor specimens taken from malignant glioma patients undergoing surgery. (Phase II) III. Tumor concentration of OSI-774 (erlotinib) and CCI-779 (temsirolimus). (Phase II)

OUTLINE: This is a multicenter, phase I, dose-escalation study of temsirolimus followed by a phase II study. Patients are stratified according to study phase (I vs II), histology at study enrollment (glioblastoma multiforme or gliosarcoma vs anaplastic glioma), preoperative candidacy (yes vs no), and presence of measurable or evaluable disease (yes vs no).

PHASE I: Patients receive oral erlotinib once daily on days 1-28 and temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of temsirolimus until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PHASE II: Patients receive temsirolimus at the MTD and erlotinib as in phase I.

PHASE II (preoperative component): Patients who are surgical candidates may opt to undergo surgical resection of the tumor. Beginning 5-7 days before surgery, these patients receive oral erlotinib once daily until surgery. Patients also receive temsirolimus IV over 30 minutes at the MTD and then undergo surgical resection of the tumor 3-24 hours later. Beginning 2-4 weeks after surgery, patients receive temsirolimus at the MTD and erlotinib as in phase I.

PROJECTED ACCRUAL: A total of 3-24 patients will be accrued for the phase I portion of the study within 1-8 months. A total of 50 patients (32 patients with glioblastoma multiforme and 18 with anaplastic glioma) will be accrued for the phase II portion of the study within 8-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven intracranial glioblastoma multiforme (GBM) or gliosarcoma (GS), anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic mixed oligoastrocytoma (AMO), or malignant astrocytoma not otherwise specified (NOS) will be eligible for this protocol; patients will be eligible if the original histology was low-grade glioma and a subsequent histological diagnosis of a malignant glioma is made
* All patients must sign an informed consent indicating that they are aware of the investigational nature of this study; patients must have signed an authorization for the release of their protected health information; patients must be registered in the Adult Brain Tumor Consortium (ABTC) Central Office database prior to treatment with study drug
* Patients must have a life expectancy > 8 weeks
* Patients must have a Karnofsky performance status of >= 60
* Patients must have recovered from the toxic effects of prior therapy: 4 weeks (28 days) from any investigational agent, 4 weeks (28 days) from prior cytotoxic therapy, two weeks (14 days) from vincristine, 6 weeks (42 days) from nitrosoureas, 3 weeks (21 days) from procarbazine administration, and 1 week (7 days) for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count); any questions related to the definition of non-cytotoxic agents should be directed to the study chair
* WBC >= 2,000/ul
* ANC >= 1,500/mm^3
* Platelet count of >= 100,000/mm^3
* Hemoglobin >= 10 gm/dl
* Total bilirubin within normal institutional limits
* AST (SGOT)/ALT (SGPT) =< 2.5 X institutional ULN
* Creatinine < 1.5 mg/dL
* Patients must have cholesterol level =< 350 mg/dl and triglycerides level =< 400 mg/dl
* Patients must have shown unequivocal evidence for tumor progression by MRI or CT scan; a scan should be performed within 14 days prior to registration; the same type of scan, i.e., MRI or CT must be used throughout the period of protocol treatment for tumor measurement
* Patients must have failed prior radiation therapy and must have an interval of greater than or equal to 6 weeks (42 days) from the completion of radiation therapy to study entry
* Patients with prior therapy that included interstitial brachytherapy or stereotactic radiosurgery must have confirmation of true progressive disease rather than radiation necrosis based upon either PET or Thallium scanning, MR spectroscopy or surgical documentation of disease
* Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply:

  * They have recovered from the effects of surgery
  * Residual disease following resection of recurrent tumor is not mandated for eligibility into the study; to best assess the extent of residual disease post-operatively, a CT/ MRI should be done no later than 96 hours in the immediate post-operative period or at least 4 weeks post-operatively, within 14 days prior to registration; if the 96-hour scan is more than 14 days before registration, the scan needs to be repeated; if the steroid dose is increased between the date of imaging and registration, a new baseline MRI/CT is required on a stable or decreasing steroid dosage for at least 5 days
* PHASE I: Patients may have had treatment for any number of prior relapses; relapse is defined as progression following initial therapy (i.e. radiation+/- chemo if that was used as initial therapy)
* PHASE I: For the baseline MRI or CT scan prior to registration, patients in the Phase I component should be on a steroid dose that has been stable for at least 5 days prior to the scan; if the steroid dose is increased between the date of imaging and registration a new baseline MR/CT is required
* PHASE II: Patients may have had treatment for no more than 2 prior relapses; relapse is defined as progression following initial therapy (i.e. radiation+/- chemo if that was used as initial therapy); the intent therefore is that patients had no more than 3 prior therapies (initial and treatment for 2 relapses); if the patient had a surgical resection for relapsed disease and no anti-cancer therapy was instituted for up to 12 weeks, and the patient undergoes another surgical resection, this is considered as 1 relapse; for patients who had prior therapy for a low-grade glioma, the surgical diagnosis of a high-grade glioma will be considered the first relapse
* PHASE II: Unstained slides or tissue blocks must be available from at least one prior surgery; if available, frozen tissue is also requested from earlier surgeries
* PHASE II: Patients who are eligible for participation in the phase II component of the study may be enrolled in a pre-operative study to evaluate biological and/or tissue correlates
* PHASE II: For the baseline MRI or CT scan prior to registration, patients in the phase II component who are not participating in the pre-operative component of the study should be on a steroid dose that has been stable for at least 5 days prior to the scan; if the steroid dose is increased between the date of imaging and registration a new baseline MR/CT is required
* PHASE II: For the patients in the preoperative component, only a scan showing progression is required; for this scan only stable steroids are not required; following surgery, a scan should be done no later than 96 hours or at least 4 weeks from surgery and on a steroid dose that is stable or decreasing; treatment with OSI-774 (erlotinib) and CCI-779 (temsirolimus) post-operatively should start no later than 14 days after the scan; if the 96-hour scan is more than 14 days before treatment is initiated, the scan needs to be repeated on a stable or decreasing steroid dose

Exclusion Criteria:

* Patients must not be on an enzyme-inducing anti-epileptic drug (EIAED); if previously on an EIAED, the patient must be off of it for at least two weeks prior to registration
* Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy
* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible
* Patients must not have active infection or serious intercurrent medical illness
* Patients must not be pregnant/breast feeding and must agree to practice adequate contraception; women of childbearing potential must have a negative B-HCG pregnancy test documented within 7 days prior to registration; patients must not be pregnant; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients must not have any disease that will obscure toxicity or dangerously alter drug metabolism
* Patients must not have received prior therapy with CCI-779 (temsirolimus), OSI-774 (erlotinib) or other mTOR or epidermal growth factor receptor inhibitors
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study due to possible retro-viral drug interactions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2005-04; Primary Completion 2010-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wen, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (8):
- United States (8):
  - University of California Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - National Cancer Institute Neuro-Oncology Branch, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- [Result] Wen PY, Chang SM, Lamborn KR, Kuhn JG, Norden AD, Cloughesy TF, Robins HI, Lieberman FS, Gilbert MR, Mehta MP, Drappatz J, Groves MD, Santagata S, Ligon AH, Yung WK, Wright JJ, Dancey J, Aldape KD, Prados MD, Ligon KL. Phase I/II study of erlotinib and temsirolimus for patients with recurrent malignant gliomas: North American Brain Tumor Consortium trial 04-02. Neuro Oncol. 2014 Apr;16(4):567-78. doi: 10.1093/neuonc/not247. Epub 2014 Jan 26. PMID 24470557

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between 2005 and 2008. Patients were recruited from outpatient medical clinics and referrals.
Groups:
- Phase I (Erlotinib & Temsirolimus): PHASE I: Oral erlotinib 1 daily days 1-28 (150mg), temsirolimus IV 30 minutes days 1, 8, 15, 22 (dose escalation). Every 28 days until disease progression or unacceptable toxicity.
  erlotinib: Given orally
  temsirolimus: Given IV
  pharmacological study: Correlative studies
- Phase II (Erlotinib & Temsirolimus): Oral erlotinib 1 daily days 1-28 (150mg), temsirolimus IV 30 minutes days 1, 8, 15, 22 at MTD phse I. Every 28 days until disease progression or unacceptable toxicity.
  PHASE II (preoperative component): Patients who are surgical candidates may opt to undergo surgical resection of the tumor. Beginning 5-7 days before surgery, these patients receive oral erlotinib once daily until surgery. Patients also receive temsirolimus IV over 30 minutes at the MTD and then undergo surgical resection of the tumor 3-24 hours later. Beginning 2-4 weeks after surgery, patients receive temsirolimus at the MTD and erlotinib as in phase I.
  therapeutic conventional surgery: Undergo surgical resection
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Phase I (Erlotinib & Temsirolimus) | Phase II (Erlotinib & Temsirolimus)
Started | 22 | 47
Completed | 21 (12 of Phase I pts treated at MTD and hence considered part of the Phase II analysis) | 47 (12 additional pts from phase 1 study were used in analysis for Phase 2 as they were treated at MTD)
Not Completed | 1 | 0
Not completed — 1 pt never had had RX due rapid decline | 1 | 0

BASELINE CHARACTERISTICS:
Population: pts had to meet eligibility criteria and recieve at least one dose of treatment.
  22 eligible pts enrolled in phase 1, but 1 pt declined before starting any treatment and was excluded from analysis - 12 pts were treated at MTD and thus included in the Phase 2 analysis, hence only 9 patients remained for analysis for phase 1
Groups:
- Phase I n=9: PHASE I: Oral erlotinib 1 daily days 1-28 (150mg), temsirolimus IV 30 minutes days 1, 8, 15, 22 (dose escalation). Every 28 days until disease progression or unacceptable toxicity.
  erlotinib: Given orally
  temsirolimus: Given IV
- Phase II n=16: Oral erlotinib 1 daily days 1-28 (150mg), temsirolimus IV 30 minutes days 1, 8, 15, 22 at MTD phse I. Every 28 days until disease progression or unacceptable toxicity.
  Anaplastic Glioma
  erlotinib: Given orally
  temsirolimus: Given IV
- Phase II n=43: Oral erlotinib 1 daily days 1-28 (150mg), temsirolimus IV 30 minutes days 1, 8, 15, 22 at MTD phse I. Every 28 days until disease progression or unacceptable toxicity.
  Glioblastoma
  erlotinib: Given orally
  temsirolimus: Given IV
- Total: Total of all reporting groups
Arm/Group | Phase I n=9 | Phase II n=16 | Phase II n=43 | Total
Number analyzed (Participants) | 9 | 16 | 43 | 68
Age, Continuous [Median (Full Range); unit: years] | 57 [33 to 74] | 47 [29 to 72] | 50 [20 to 69] | 51 [20 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 12 | 20
  Male | 5 | 12 | 31 | 48
Karnofsky Performance Scale (KPS) [Median (Full Range); unit: units on a scale] — The KPS scores range from 0 (lowest score) to 100 (highest score).
  The higher the score the better able to carry out daily activities
  100-80: able to carry on normal activity and to work; No special care
  70-50: Unable to work; able to live at home and care for most personal needs; varying amount of assistance needed
  40-10: unable to care for self, requires equivalent of institutional or hospital care; diseases may be progressing rapidly
  0: dead
  units on a scale | 90 [70 to 100] | 90 [60 to 100] | 90 [60 to 100] | 90 [60 to 100]
Prior Chemotherapy treatments [Median (Full Range); unit: treatments] | 2 [0 to 3] | 1 [1 to 3] | 1 [0 to 3] | 1 [0 to 3]
Histology [Number; unit: participants]
  anaplastic glioma | 3 | 16 | 0 | 19
  glioblastoma | 6 | 0 | 43 | 49

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (Phase I)
Description: Oral erlotinab at 150mg constant dose, 3 pts will be treated with temsirolimus IV with escalating doses, starting at 50mg. Doses will increase or decrease based on toxicity observed.
  3 pts will be treated at each dose level - 3 dose levels were observed: 50mg, 25mg, and 15mg
Time Frame: based on first 4 weeks of treatment - cycle 1
Population: Per protocol -
Measure: Number; unit: mg
Groups:
- Phase I - Dose Escalation: Oral erlotinib 1 daily days 1-28 (150mg), temsirolimus IV 30 minutes days 1, 8, 15, 22 at (dose escalation or dose de-escalation). Every 28 days until disease progression or unacceptable toxicity.
  Dose levels: cohort 1 - 50mg - 3pts cohort 2 - 25mg -6pt cohort 3 - 15mg - 12pts
Arm/Group | Phase I - Dose Escalation
Number analyzed (Participants) | 21
mg | 15

2. Primary Outcome: Safety/Dose Limiting Toxities Phase I
Description: Dose limiting toxities defined as: grade 3 thrombocytopenia, grade 4 anemia and neutropenia, grade >/= nonhematologic toxicity, and failure to recover from toxicites to be eligible for retreatment in 2 weeks of the last dose of either drug. Also grade 3 nonhematologic toxicities only if they wre refractory to maxiaml medical therapy.
  MTD defined as dose at which fewer than one-third of patients experienced a DLT
  Outcome measure defines number of participants who had a defined dose limiting toxicity.
Time Frame: first 4 weeks of treatment
Measure: Number; unit: participants
Groups:
- Phase 1 - 50mg: Oral erlotinib 1 daily days 1-28 (150mg), temsirolimus IV 30 minutes days 1, 8, 15, 22 (50mg). Every 28 days until disease progression or unacceptable toxicity.
- Phase 1 - 25 mg: Oral erlotinib 1 daily days 1-28 (150mg), temsirolimus IV 30 minutes days 1, 8, 15, 22 (25mg). Every 28 days until disease progression or unacceptable toxicity.
- Phase 1 - 15mg: PHASE I: Oral erlotinib 1 daily days 1-28 (150mg), temsirolimus IV 30 minutes days 1, 8, 15, 22 (15mg). Every 28 days until disease progression or unacceptable toxicity.
Arm/Group | Phase 1 - 50mg | Phase 1 - 25 mg | Phase 1 - 15mg
Number analyzed (Participants) | 3 | 6 | 12
participants | 2 | 3 | 3

3. Primary Outcome: Efficacy - Response Phase 1
Description: pt must have at least 8 weeks of treatment to receive MRI scan, scans are every other cycle (every 2 months). Response measured by a bidimensionally measured leison and clearly defined margins by CT or MRI scan.
  Complete Response (CR): complete disappearance of all measurable and evaluable disease. No new lesions, not on any steroids Partial Response (PR): >= 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesions. No progression of evaluable disease. No new lesions. Steriod dose must be no greater than max used in 1st 8wks of therapy Stable: not qualify for CR, PR, or progression. Steriod dose must be no greater than max used in 1st 8wks of therapy Progression (PD): 25% increase in the sum of products of all measurable lesions over smallest sum observed, OR clear worsening or failure to return for evalution due to death or deteriorating condition (unless clearly unrelated to brain cancer).
Time Frame: at least 8 weeks of treatment
Population: Response was reviewed only in those patients treated at the MTD (15mg temsirolimus)
Measure: Number; unit: participants
Groups:
- Phase I 15mg Temsirolimus (MTD Dose): PHASE I: Oral erlotinib 1 daily days 1-28 (150mg), temsirolimus IV 30 minutes days 1, 8, 15, 22 (15mg). Every 28 days until disease progression or unacceptable toxicity.
  erlotinib: Given orally
  temsirolimus: Given IV
Arm/Group | Phase I 15mg Temsirolimus (MTD Dose)
Number analyzed (Participants) | 12
participants
  Complete Response | 0
  Partial response | 1
  Stable | 2
  Progressive Disease | 9

4. Primary Outcome: Pharmacokinetics (Phase I)
Description: Tersirolimus Cmax (ng/mL) for cycle 1 is presented in the outcome measure table below for the 3 dose levels
  blood samples (5ml) was collected in EDTA containing tubes on days 1 and 2 of cycle 1
  Collection time points: prior to dosing of both drugs, at end of temsirolimus infusion and at 1,2,4,6, and 24 hr after erlotinib administration
Time Frame: Days 1, 2 of cycle 1, prior to dosing of both drugs, at end of temsirolimus infusion and at 1,2,4,6, and 24 hr after erlotinib administration
Population: per protocol
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1 - 15mg | Phase 1 - 25 mg | Phase 1 - 50mg
Number analyzed (Participants) | 11 | 6 | 3
ng/mL | 460 (219) | 428 (115) | 451 (281)

5. Primary Outcome: Progression-free Survival at 6 Months (Phase II)
Description: Progression (PD): 25% increase in the sum of products of all measurable lesions over smallest sum observed, OR clear worsening or failure to return for evalution due to death or deteriorating condition (unless clearly unrelated to brain cancer).
  Responses had to be present on 2 consecutive scans and were centrally reviewed.
Time Frame: Evaluated at baseline and every other cycle, till Month 6
Population: Primary endpoint PFS6 date of registration; Sample size chosen to discriminate between 15% & 35% PFS6 rates for GBM patients. With accrual 32 GBM patients, trial would be considered successful if 8 achieved PFS6. This yields 0.92 power to detect a 35% PFS6 rate, with 0.90 probability of rejecting the treatment regimen if the PFS6 rate is only 15%.
Measure: Number; unit: participants
Arm/Group | Phase II n=43
Number analyzed (Participants) | 43
participants | 6

ADVERSE EVENTS:
Time Frame: Adverse Events were collected weekly for the first cycle and then at the start of each cycle while on treatment and at time of off study.
Groups:
- Phase II (Erlotinib & Erlotinib): Oral erlotinib 1 daily days 1-28 (150mg), temsirolimus IV 30 minutes days 1, 8, 15, 22 at MTD phse I. Every 28 days until disease progression or unacceptable toxicity.
  PHASE II (preoperative component): Patients who are surgical candidates may opt to undergo surgical resection of the tumor. Beginning 5-7 days before surgery, these patients receive oral erlotinib once daily until surgery. Patients also receive temsirolimus IV over 30 minutes at the MTD and then undergo surgical resection of the tumor 3-24 hours later. Beginning 2-4 weeks after surgery, patients receive temsirolimus at the MTD and erlotinib as in phase I.
  therapeutic conventional surgery: Undergo surgical resection
  laboratory biomarker analysis: Correlative studies
Arm/Group | Phase I (Erlotinib & Temsirolimus) | Phase II (Erlotinib & Erlotinib)
Serious Adverse Events (participants affected / at risk) | 3/21 | 2/59
Other Adverse Events (participants affected / at risk) | 21/21 | 37/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (Erlotinib & Temsirolimus) (N=21) | Phase II (Erlotinib & Erlotinib) (N=59)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) — Cardiac ischemia
fever (General disorders) | 1 (1) | 0 (0)
generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — normal ANC
retinopathy (Eye disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (Erlotinib & Temsirolimus) (N=21) | Phase II (Erlotinib & Erlotinib) (N=59)
White blood Cells (Investigations) | 2 (2) | 0 (0) — Leukopenia
Platelets (Investigations) | 4 (4) | 2 (2) — Thrombocytopenia
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
fatigue (General disorders) | 2 (2) | 2 (2)
hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
hypophosphatemia (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
hypotension (Cardiac disorders) | 2 (2) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Liver Function Test abnormality (Investigations) | 3 (3) | 1 (1) — SGOT, SGPT
Mucositis oral (Gastrointestinal disorders) | 6 (6) | 5 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 8 (8) | 10 (10)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lymphocyte count decrease (Investigations) | 0 (0) | 5 (5) — lymphopenia
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Pain in Limb

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less